CLINICAL TRIAL: NCT01675076
Title: A Randomized Controlled Trial to Investigate Whether a Strategy of Continued Versus Interrupted Novel Oral Anti-coagulant at the Time of Device Surgery, in Patients With Moderate to High Risk of Arterial Thrombo-embolic Events, Leads to a Reduction in the Incidence of Clinically Significant Hematoma
Brief Title: Strategy of Continued Versus Interrupted Novel Oral Anti-coagulant at Time of Device Surgery in Patients With Moderate to High Risk of Arterial Thromboembolic Events
Acronym: BRUISECONTROL2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Boehringer Ingelheim (Industry); Heart and Stroke Foundation of Canada (Other); Bayer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOHI-05
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Hematoma
Keywords: Hematoma; novel oral anti-coagulant (NOAC); Device surgery
MeSH Terms: conditions — Hematoma | interventions — Dabigatran; Rivaroxaban; apixaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continued NOAC (Experimental): - Patients continue on their chronic dose of Dabigatran or Rivaroxaban or Apixaban throughout
  Interventions: Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban
- Interrupted NOAC (Active Comparator): Interrupted Dabigatran:
  * Discontinue Dabigatran 1 day before surgery if GFR > 50 mL/min or discontinue 2 days before surgery if GFR 30-50 mL/min
  * Resume Dabigatran at next regular dose timing >or = 24 hours after the end of surgery
  Interrupted Rivaroxaban:
  * Discontinue Rivaroxaban 1 full day before surgery
  * Resume Rivaroxaban at next regular dose timing >or = 24 hours after the end of surgery
  Interrupted Apixaban:
  * Discontinue Apixaban 1 full day before surgery
  * Resume Apixaban at next regular dose timing >or = 24 hours after the end of surgery
  Interventions: Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban

INTERVENTIONS:
Drug: Dabigatran — NOAC
  Other Names: Pradaxa
Drug: Rivaroxaban — NOAC
  Other Names: Xarelto
Drug: Apixaban — NOAC
  Other Names: Eliquis

SUMMARY:
The purpose of this study is to determine the best strategy to manage novel oral anti-coagulants (NOACs) at the time of pacemaker or defibrillator surgery. The Investigators hypothesize that performing device surgery without interruption of the novel oral anti-coagulant will result in a reduced rate of clinically significant hematoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized trial, with 1:1 randomization to either continued NOAC or interrupted NOAC in patients with non-rheumatic atrial fibrillation or atrial flutter and at moderate to high risk of arterial thrombo-embolic events who require device surgery.

All patients in the study will be receiving Dabigatran or Rivaroxaban or Apixaban for at least 5 days prior to enrollment. The peri-operative management of the NOAC the patient is receiving is randomized to Interrupted NOAC or Continued NOAC.

Interrupted NOAC arm:

1. Interrupted Dabigatran

   * based on renal function, patients will discontinue Dabigatran 1 day before surgery if GFR > 50 mL/min, and 2 days before surgery if GFR is 30-50 mL/min.
   * Dabigatran will be resumed at the next regular dose time, > or = 24 hours after the end of surgery.
2. Interrupted Rivaroxaban

   * patients will discontinue Rivaroxaban 1 full day before surgery.
   * Rivaroxaban will be resumed at the next regular dose time, > or = 24 hours after the end of surgery.
3. Interrupted Apixaban

   * patients will discontinue Apixaban 1 full day before surgery.
   * Apixaban will be resumed at the next regular dose time, > or = 24 hours after the end of surgery.

Continued NOAC arm:

-patients will continue their chronic dose of Dabigatran or Rivaroxaban or Apixaban throughout.

All patients will have a baseline clinical lab test of serum creatinine or GRF measured.

Patients will be seen post-op on the day of their surgery for assessment of the surgical site and each day throughout their hospital stay by a blinded member of the research team. A telephone follow-up will be done on day 3-4 post surgery by an unblinded team member. All patients are seen 1-2 weeks post-op at their first routine post-op device clinic visit, for surgical site assessment by the blinded assessor and to complete Quality of Life questionnaires. Patients will be seen for assessment in the case of any bleeding or development of pocket swelling or hematoma. Patients developing a hematoma will be followed until resolution of the hematoma.

ELIGIBILITY:
Inclusion Criteria:

* any patient undergoing device surgery (ie. de novo device implant or pulse generator change or lead replacement or pocket revision)
* receiving Dabigatran or Rivaroxaban or Apixaban for at least 5 days prior to enrollment
* non-rheumatic atrial fibrillation and/or atrial flutter at moderate or high risk of ATE defined as: i) CHA2DS2VASc score greater than or equal to 2 OR ii) CHA2DS2VASc score < 2 with plan for cardioversion or defibrillation threshold testing at time of device surgery

Exclusion Criteria:

* unable or unwilling to provide informed consent
* history of noncompliance of medical therapy
* active device infection
* eGFR < 30 mL/min
* contraindication to NOAC
* rheumatic valvular disease with hemodynamically significant valve lesion
* mechanical heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Clinically significant hematoma | 2 weeks post-op or until resolution of hematoma
  Defined as:
  1. Hematoma requiring re-operation
     - Defined as a hematoma that continues to expand despite all appropriate non-operative measures, or is producing impending or actual wound breakdown or skin necrosis. Minor hematomas that are evacuated at the time of other re-operation (eg. for lead repositioning) are not considered as a primary outcome.
     or
  2. Hematoma resulting in prolongation of hospitalization
     - Defined as extended hospitalization or rehospitalization for > 24 hours, post index surgery, primarily due to hematoma.
     or
  3. Hematoma requiring interruption of anti-coagulation. - Defined as reversal or intentional withholding of all anticoagulation for > or = 24 hours, in response to wound hematoma.

SECONDARY OUTCOMES:
Composite of major peri-operative bleeding events and thrombo-embolic events | 2 weeks post-op
  1. Each of the components of the primary outcome
  2. Composite of all other major peri-operative bleeding events defined as:
     * hemothorax
     * cardiac tamponade
     * significant pericardial effusion
  3. Thrombo-embolic events defined as:
     * transient ischemic attack
     * stroke
     * deep venous thrombosis
     * pulmonary embolism
     * peripheral embolus to limb
     * peripheral embolus to other major organ
  4. All cause mortality
  5. Cost utilization
  6. Patient quality of life and peri-operative pain, and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Vidal Essebag, MD, Principal Investigator — McGill University; Jeff Healey, MD, Study Chair — McMaster University
Locations (15):
- Canada (14):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta-ECAT Group, Edmonton, Alberta
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Hamilton Health Sciences General Campus, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Rouge Valley Health System-Centenary Campus, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Hotel Dieu, Montreal, Quebec
  - McGill University Health Centre/Montreal General Hospital, Montreal, Quebec
  - Hopital Sacre-Coeur, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Hopital Fleurimont, Sherbrooke, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Galilee Medical Center, Nahariya, Israel

REFERENCES:
- [Result] Birnie DH, Healey JS, Wells GA, Ayala-Paredes F, Coutu B, Sumner GL, Becker G, Verma A, Philippon F, Kalfon E, Eikelboom J, Sandhu RK, Nery PB, Lellouche N, Connolly SJ, Sapp J, Essebag V. Continued vs. interrupted direct oral anticoagulants at the time of device surgery, in patients with moderate to high risk of arterial thrombo-embolic events (BRUISE CONTROL-2). Eur Heart J. 2018 Nov 21;39(44):3973-3979. doi: 10.1093/eurheartj/ehy413. PMID 30462279
- [Derived] Essebag V, Healey JS, Joza J, Nery PB, Kalfon E, Leiria TLL, Verma A, Ayala-Paredes F, Coutu B, Sumner GL, Becker G, Philippon F, Eikelboom J, Sandhu RK, Sapp J, Leather R, Yung D, Thibault B, Simpson CS, Ahmad K, Toal S, Sturmer M, Kavanagh K, Crystal E, Wells GA, Krahn AD, Birnie DH. Effect of Direct Oral Anticoagulants, Warfarin, and Antiplatelet Agents on Risk of Device Pocket Hematoma: Combined Analysis of BRUISE CONTROL 1 and 2. Circ Arrhythm Electrophysiol. 2019 Oct;12(10):e007545. doi: 10.1161/CIRCEP.119.007545. Epub 2019 Oct 15. PMID 31610718